CLINICAL TRIAL: NCT04502212
Title: An Open-Label, Pilot Study to Assess the Effects of Hepatic Ultrasound Insonification on Glucometabolic Parameters in Subjects With T2DM
Brief Title: Pilot Study to Assess the Effects of Hepatic Ultrasound Insonification on Subjects With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Electric Research (Industry)
Collaborators: ProSciento, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GE Research HUI-01
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Insonification (Experimental): All subjects enrolled will receive a 3-day, 15 minute per day ultrasound insonification targeting the portis hepatis (liver).
  Interventions: Device: Hepatic Ultrasound Insonification

INTERVENTIONS:
Device: Hepatic Ultrasound Insonification — Hepatic ultrasound insonification will be performed after an overnight fast (no food or drinks except for water for at least 10 hours) at approximately the same time on each day for three days.

SUMMARY:
This research study is being done to evaluate the effect of hepatic ultrasound insonification on whole-body insulin sensitivity and evaluate the safety and tolerability of hepatic ultrasound insonification in subjects with Type 2 Diabetes Mellitus (T2DM). "Insonify/insonification" is defined as applying to an area or an object carefully-controlled sound waves, typically as in ultrasound imaging. GE Research is sponsoring this research study. The purpose of this research study is to:

* Evaluate the effect of liver ultrasound waves on changes from baseline in whole-body insulin sensitivity
* Test the safety and tolerability of liver ultrasound waves in subjects with Type 2 Diabetes Mellitus
* Evaluate the effect of liver ultrasound waves on change from baseline in glucose tolerance and insulin secretion
* Evaluate the effect of liver ultrasound waves on glucose metabolism

Insulin sensitivity refers to how sensitive the body's cells are in response to insulin.

Glucose tolerance refers to the body's ability to handle (tolerate) glucose. Insulin secretion is a process in which the body releases insulin in response to glucose levels in the blood becoming elevated.

The study device used in this study is cleared for use by the United States Food and Drug Administration (FDA) for ultrasound diagnostic exams, however it has not been tested or approved specifically for modulation of metabolism in people with diabetes. The use of the study device in this study is investigational and is considered a Non-Significant Risk (NSR).

DETAILED DESCRIPTION:
This was an open label, exploratory pilot study to assess the effects of hepatic ultrasound insonification on glucometabolic parameters in subjects with T2DM through selective hepatic ultrasound of the porta hepatis region of the liver utilizing pulsed ultrasound. The study was to consist of 1 cohort comprising up to 15 subjects. Dropouts and withdrawals could have been replaced until the anticipated number of subjects completed the study. Finally, the study consisted of one cohort with 36 subjects enrolled, including 20 screen failures, 15 subjects that completed the study (1 completer had an incorrect infusion parameter and was removed from clamp analysis), and 1 subject that was discontinued at the discretion of the Investigator. As this was an exploratory, open-label study, no randomization or blinding was performed and no-unblinding codes were required.

The study included a Screening Period, Observational Period 1, 3 consecutive days of hepatic ultrasound insonification, and Observational Period 2. Each Observational Period was divided into an In-house Period and an Outpatient Visit (OPV). The Screening Period was performed up to 28 days prior to the first In-house Period. For eligible subjects with a body mass index (BMI) > 35.0 and ≤ 40.0 kg/m2 and/or a waist circumference > 40 and ≤ 45 inches, an ultrasound examination was added to confirm eligibility, and the Screening Period was extended to at least 30 days. The first Observational Period lasted approximately 2-weeks (Days -1 to 14). On the morning of Day -1, subjects checked into the clinic for a 3-day In-house Period; subjects may have been released from the clinic on Day 2. Subjects were contacted via telephone every other day until the next In-house Period. On Day 8, subjects checked into the clinic for an OPV. On Day 15, subjects checked into the clinic in fasting conditions for a 4-day In-house Period. Insonifications were performed on three consecutive days (Days 15, 16 and 17). Subjects may have been released from the clinic on Day 18. The second Observational Period lasted 11 days (Days 18 to 28). Subjects were contacted via telephone every other day until the Follow-up Visit. On Day 22, subjects checked into the clinic for the OPV. The Follow-up Visit was performed on Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with type 2 diabetes ≥ 12 months.
2. Age ≥ 21 and ≤ 75 years.
3. Stable treatment with diet and exercise or stable treatment with metformin monotherapy. Stable treatment is defined as no change in treatment during the last 3 months.
4. HbA1c > 6.5% and< 10% by local laboratory analysis (one retest is permitted with the result of the last test being conclusive).
5. Body Mass Index (BMI) ≥ 18 to ≤ 35.0 kg/m2.
6. Waist circumference ≤ 40 inches (≤ 102 cm).
7. Considered generally healthy upon completion of medical history, physical examination and biochemical investigations as judged by the Principal Investigator.
8. Female subjects must be non-pregnant and non-lactating and have a negative serum pregnancy test at Screening. Females may be surgically sterile, postmenopausal or of child-bearing potential. Females of childbearing potential must be using an acceptable method of birth control.
9. Ability to provide written informed consent.

Exclusion Criteria:

1. History or current diagnosis with T1DM or T2DM subjects on insulin or other injectable therapies not allowed for this study (as listed in table of Prohibited Medication below).
2. A subject who is already indicated for medication escalation of their current diabetic therapy, or, who based upon study entry criteria, would be indicated for medication escalation during the course of the study (as assessed by the qualified Principal Investigator).
3. A subject who has diabetic complications, i.e., acute proliferative retinopathy or maculopathy, severe gastroparesis, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Principal Investigator.
4. Recurrent severe hypoglycemia (more than 1 event ≤ 6 month) or hypoglycemic unawareness or recent severe ketoacidosis (hospitalization ≤ 6 month), as judged by the Principal Investigator.
5. Persistent systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 95 mm Hg at screening. (Subjects may be re-checked once on the same day).
6. Treatment with antihypertensive medication is not allowed, unless antihypertensive medication is given on a stable dose for at least 2 months prior to screening.
7. Subjects with a clinically significant history or active disease of any of the following body systems: pulmonary, neurological (including dementia, neurodegenerative disease, movement disorder, spinal disorders), pancreatic (including pancreatitis), immunological or systemic inflammatory (including systemic lupus erythematosus [SLE], rheumatoid arthritis [RA]), dermatological, endocrine, genitourinary or hematological (including sickle cell anemia or other anemia syndromes, monocytosis, thrombocytopenia).
8. Subjects with a history or clinically active malignancy (history of basal cell carcinoma [BCC] is allowed).
9. History or current diagnosis of cardiac dysrhythmias or heart disease, defined as symptomatic heart failure (New York Heart Association class III or IV), myocardial infarction, unstable angina requiring medication.
10. Transient ischemic attack [TIA], cerebral infarct, or cerebral hemorrhage.
11. Invasive cardiovascular procedure, such as coronary artery bypass graft surgery (CABG), or angioplasty/percutaneous coronary intervention (PCI) within 6 months of screening.
12. PHistory of or presence of clinically significant ECG findings (e.g., QTcF > 450 msec for males, QTcF > 470 msec for females, LBBB) at Screening, or cardiac arrhythmia requiring medical or surgical treatment within 6 months prior to screening.
13. History of renal disease or abnormal kidney function tests at Screening (glomerular filtration rate [GFR] < 60 mL/min/1.73m2 as estimated using the MDRD equation).
14. History or clinically significant active hepatic disease or clinically significant abnormal hepatic function tests at Screening suggestive of hepatic impairment (e.g., ALT and/or AST >2 x ULN), total bilirubin > 1 x ULN).
15. Subjects with a history or presence of any psychiatric disorder that, in the opinion of the Principal Investigator, might confound the results of the trial or pose additional risk in administering the investigational product to the subject.
16. Personal or family history of hypercoagulability or thromboembolic disease, including deep vein thrombosis and/or pulmonary embolism (PE)
17. History of surgical treatment for obesity (bariatric surgery, gastric banding, etc.) or any other gastrointestinal surgery (including appendectomy, cholecystectomy), any malabsorption disorder, severe gastroparesis, any GI procedure for weight loss (including LAP-BAND®), as well as clinically significant gastrointestinal disorders (e.g. peptic ulcers, severe GERD) at Screening.
18. History of any major surgery within 3 months prior to screening.
19. Any nerve stimulation study or implanted stimulator, including previously or currently implanted vagus nerve stimulator, previously or currently implanted spinal cord stimulator, other implanted electronic medical device, such as implanted pacemaker or cardioverter/defibrillator (AICD) or history of seizures.
20. Diagnosis of sleep apnea.
21. Participation in an investigational study within 30 days of screening or 5 half-lives within the last dose of any investigational product given during the investigational study, whichever is longer.
22. Current use of any drugs (other than current treatment for diabetes mellitus) that are known to interfere with glucose or insulin metabolism as stated below in table prohibited medication.
23. Thyroid hormone use is not allowed unless medication is given on a stable dose for at least 3 months prior to screening.
24. Chronic use of acetaminophen, and inability to wash-out and abstain from use during the study, as it would interfere with the CGMS assessment.
25. Subject is unable to tolerate adhesive tape or has any unresolved adverse skin reaction in the area of the sensor placement.
26. Implanted pacemaker or cardioverter/defibrillator (AICD).
27. Daily use of more than 5 cigarettes/day or equivalent use of any tobacco- or nicotine-containing product (such as, but not limited to vaping, transdermal nicotine patch, nicotine gum use, etc.) within 4 weeks prior to screening. Subjects must be able to abstain from any tobacco or nicotine containing products during confinement period.
28. Any use of marijuana within 4 weeks prior to screening and positive test at screening.
29. History of any active infection, except mild viral disease, such as common cold, within 30 days prior to screening.
30. History of any recent traumatic injury, including intracerebral hemorrhage and visceral injury.
31. History of alcohol or illicit drug abuse as judged by the Principal Investigator within past 12 months or positive test at screening. Any use of alcohol within 4 days prior to baseline assessment. Subjects must be able to abstain from any alcohol during confinement period.
32. Known history or positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), human immunodeficiency virus type 1 (HIV-1) or type 2 (HIV-2)
33. Donation or loss of > 500 mL of blood or blood product within 56 days prior to screening
34. Mental incapacity, unwillingness or language barriers precluding adequate understanding and to follow verbal commands during the ultrasound session or cooperation.
35. An abdominal ultrasound scan or exam within 1 month prior to screening and/or any pre-planned ultrasound examinations during the study, or the need to participate in any unplanned outside ultrasound procedures during study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bridgette Boggess Franey, MD, Principal Investigator — ProSciento, Inc.
Locations (1):
- ProSciento, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy JC, Matthews DR, Hermans MP. Correct homeostasis model assessment (HOMA) evaluation uses the computer program. Diabetes Care. 1998 Dec;21(12):2191-2. doi: 10.2337/diacare.21.12.2191. No abstract available. PMID 9839117
- See also: Related Info — https://www.dtu.ox.ac.uk/homacalculator/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 36 subjects enrolled into the screening visit, 16 subjects were enrolled into the study and 14 subjects completed the study for all outcomes. Of the 16 subjects enrolled, 1 subject discontinued the study at the discretion of the Investigator and 1 subject failed to complete only the clamp outcomes (i.e. completed all non-clamp outcomes) due to a clamp protocol deviation.
  Of the 16 subjects enrolled, 3 subjects failed the initial screen and were rescreened at a later date.
Groups:
- Ultrasound Insonification Effect Population: The Ultrasound Insonification Effect Population was to consist of all subjects who received at least 1 hepatic ultrasound insonification and included 14 subjects.
  The Safety Population was to consist of all subjects who received at least 1 hepatic ultrasound insonification and included 16 subjects.
  One subject had unevaluable data and was excluded from the Ultrasound Insonification Effect Population; however, the subject was included in the Safety Population.
  One subject had Step 1 of the Day 17 clamp extended by 60 minutes, per PI discretion, following a protocol deviation and was excluded from the Ultrasound Insonification Effect Population; however, the subject was included in the Safety Population.
Period: Overall Study
Arm/Group | Ultrasound Insonification Effect Population
Started | 16
Completed | 14
Not Completed | 2
Not completed — Unevaluable data; excluded from Ultrasound Insonification Effect Pop; included in Safety Pop | 1
Not completed — Clamp protocol deviation; excluded from Ultrasound Insonification Effect Pop; included in Safety Pop | 1

BASELINE CHARACTERISTICS:
Population: Demographic characteristics by subject for all enrolled subjects.
Groups:
- Ultrasound Insonification Effect Population: The Ultrasound Insonification Effect Population was to consist of all subjects who received at least 1 hepatic ultrasound insonification and completed the study for all outcomes (without being discontinued from the study at the discretion of the Investigator or failing to complete the clamp outcomes due to protocol deviation) and included 14 subjects.
  The Safety Population was to consist of all subjects who received at least 1 hepatic ultrasound insonification and included 16 subjects.
Arm/Group | Ultrasound Insonification Effect Population
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (5.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 12
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glucose Disposal Rate: Insulin Ratio During Steady State (M/I)
Description: To evaluate the effect of hepatic ultrasound insonification on changes from baseline in whole-body insulin sensitivity during a two-step hyperinsulinemic, euglycemic clamp with stable isotope labeled glucose tracer
Time Frame: Day 2 (Baseline) to Day 17
Measure: Mean (Standard Deviation); unit: mg/kg/min per microU/ml
Groups:
- Ultrasound Insonification Effect Population: The Ultrasound Insonification Effect Population was to consist of all subjects who received at least 1 hepatic ultrasound insonification and included 14 subjects.
  The Safety Population was to consist of all subjects who received at least 1 hepatic ultrasound insonification and included 16 subjects.
Arm/Group | Ultrasound Insonification Effect Population
Number analyzed (Participants) | 14
mg/kg/min per microU/ml
  Clamp Timepoint with Low Rate Insulin Infusion (Step 1) | 0.055 (0.0932)
  Clamp Timepoint with High Rate Insulin Infusion (Step 2) | 0.004 (0.0161)

2. Primary Outcome: Change From Baseline in Endogenous Glucose Production (EGP)
Description: as for outcome 1
Time Frame: Day 2 (Baseline) to Day 17
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Ultrasound Insonification Effect Population
Number analyzed (Participants) | 14
mg/kg/min
  Clamp Timepoint prior to Insulin Infusion (Fasting) | -0.004 (0.2316)
  Clamp Timepoint with Low Rate Insulin Infusion (Step 1) | -0.169 (0.4849)

3. Primary Outcome: Change From Baseline in Insulin-Mediated EGP Suppression During the Clamp Timepoint With Low Rate Insulin Infusion (Step 1)
Description: To evaluate the effect of hepatic ultrasound insonification on changes from baseline in whole-body insulin sensitivity during a two-step hyperinsulinemic, euglycemic clamp with stable isotope labeled glucose tracer
  For each clamp, the degree of EGP suppression from the fasting EGP value was to be determined during the last 30 minutes point during each step of the two-step H-E clamp using the following equation:
  % EGP suppression = 1 - (EGP clamp/EGP fasting) Partial suppression of EGP during Step 1 was to be assessed to determine hepatic insulin sensitivity and EGP suppression during Step 2 was to be measured to confirm that EGP was (near) fully suppressed to allow the determination of extrahepatic insulin sensitivity.
Time Frame: Day 2 (Baseline) to Day 17
Measure: Mean (Standard Deviation); unit: percent suppression
Arm/Group | Ultrasound Insonification Effect Population
Number analyzed (Participants) | 14
percent suppression | 10.06 (25.294)

4. Primary Outcome: Change From Baseline in Rate of Glucose Disappearance (Rd)
Description: as for outcome 1
Time Frame: Day 2 (Baseline) to Day 17
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Ultrasound Insonification Effect Population
Number analyzed (Participants) | 14
mg/kg/min
  Clamp Timepoint prior to Insulin Infusion (Fasting) | -0.004 (0.2316)
  Clamp Timepoint with Low Rate Insulin Infusion (Step 1) | 0.663 (1.6645)
  Clamp Timepoint with High Rate Insulin Infusion (Step 2) | 1.029 (3.2130)

5. Secondary Outcome: Incidence of Adverse Device Effects (ADEs) With a Severity Score of 1: Treatment Emergent Adverse Events (TEAEs) by System Organ Class and Preferred Term
Description: To evaluate safety and tolerability of hepatic ultrasound insonification in subjects with T2DM. Incidence of adverse device effects included observations of Incidence and severity of clinically significant laboratory abnormalities, Change from baseline in vital signs (blood pressure, temperature, respiratory rate, and heart rate), Incidence and severity of clinical findings on physical examination, Change from baseline in 12-lead electrocardiogram (ECG) parameters; the primary ECG endpoint was QTcF.
  To evaluate safety and tolerability of hepatic ultrasound insonification in subjects with T2DM: [Severity Score: 1=Mild; 2=Moderate; 3=Severe; 4=Life-Threatening; 5=Death]
Time Frame: Screening to Day 28
Measure: Count of Participants; unit: Participants
Groups:
- Safety Population: The Safety Population was to consist of all subjects who received at least 1 hepatic ultrasound insonification and included 16 subjects.
  The Ultrasound Insonification Effect Population was to consist of all subjects who received at least 1 hepatic ultrasound insonification and included 14 subjects.
Arm/Group | Safety Population
Number analyzed (Participants) | 16
Participants
  Subjects with at least one Treatment Emergent Adverse Event (TEAE) | 7
  Skin and subcutaneous tissue disorders | 3
  Ecchymosis | 2
  Erythema | 1
  Gastrointestinal disorders | 2
  Abdominal pain | 1
  Dyspepsia | 1
  Vomiting | 1
  General disorders and administration site conditions | 2
  Infusion site hemorrhage | 1
  Vessel puncture site swelling | 1
  Metabolism and nutrition disorders | 1
  Hypoglycaemia | 1
  Nervous system disorders | 1
  Dizziness | 1
  Vascular disorders | 1
  Thrombophlebitis | 1
  Treatment Emergent Adverse Device Effect (TEADE) | 0
  TEADE Related to Study Procedure | 0
  Serious TEADE | 0
  TEADE Leading to Study Discontinuation | 0
  Unanticipated Adverse Device Effect (UADE) | 0

6. Secondary Outcome: Incidence of Clinically Significant Laboratory Abnormalities
Description: To evaluate safety and tolerability of hepatic ultrasound insonification in subjects with T2DM
Time Frame: Screening to Day 28
Measure: Number; unit: clinically significant lab abnormalities
Arm/Group | Safety Population
Number analyzed (Participants) | 16
clinically significant lab abnormalities
  Number of Clinically Significant Lab Abnormalities | 0
  Number of Clinically Significant Changes in Hematology Laboratory Values | 0
  Number of Clinically Significant Changes in Hepatic Function Laboratory Values | 0
  Number of Clinically Significant Changes in Renal Function Laboratory Values | 0
  Number of Clinically Significant Changes in Urinalysis Laboratory Values | 0

7. Secondary Outcome: Incidence of Significant Clinical Findings on Physical Examination
Description: To evaluate safety and tolerability of hepatic ultrasound insonification in subjects with T2DM
Time Frame: Screening to Day 28
Measure: Number; unit: clinically significant phys exam finding
Arm/Group | Safety Population
Number analyzed (Participants) | 16
clinically significant phys exam finding | 0

8. Secondary Outcome: Change From Baseline in Vital Signs: Blood Pressure
Description: To evaluate safety and tolerability of hepatic ultrasound insonification in subjects with T2DM
Time Frame: Baseline to Day 28 - Baseline was defined as the last non-missing value collected prior to the first on study hepatic ultrasound insonification
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Safety Population
Number analyzed (Participants) | 16
mmHg
  Change from Baseline in Systolic Blood Pressure | -3.4 (10.89)
  Change from Baseline in Diastolic Blood Pressure | -3.0 (5.06)

9. Secondary Outcome: Change From Baseline in Vital Signs: Pulse Rate
Description: To evaluate safety and tolerability of hepatic ultrasound insonification in subjects with T2DM
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Safety Population
Number analyzed (Participants) | 16
beats/minute | -1.9 (10.62)

10. Secondary Outcome: Change From Baseline in Vital Signs: Respiratory Rate
Description: To evaluate safety and tolerability of hepatic ultrasound insonification in subjects with T2DM
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Safety Population
Number analyzed (Participants) | 16
breaths/minute | -1.0 (2.28)

11. Secondary Outcome: Change From Baseline in Vital Signs: Temperature
Description: To evaluate safety and tolerability of hepatic ultrasound insonification in subjects with T2DM
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Safety Population
Number analyzed (Participants) | 16
degrees C | 0.07 (0.531)

12. Secondary Outcome: Incidence of Clinically Significant Changes in Vital Sign Values
Description: To evaluate safety and tolerability of hepatic ultrasound insonification in subjects with T2DM
Time Frame: Screening to Day 28
Measure: Mean (Standard Deviation); unit: clinically significant changes
Arm/Group | Safety Population
Number analyzed (Participants) | 16
clinically significant changes | 0 (0)

13. Secondary Outcome: Change From Baseline in 12-lead Electrocardiogram (ECG) Parameters
Description: To evaluate safety and tolerability of hepatic ultrasound insonification in subjects with T2DM
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Safety Population
Number analyzed (Participants) | 16
msec
  Change from Baseline in QT Interval | 4.6 (20.84)
  Change from Baseline in PR Interval | -1.8 (15.26)
  Change from Baseline in QRS Interval | 1.1 (6.01)
  Change from Baseline in RR Interval | 12.4 (99.99)
  Change from Baseline in QTcF Interval | 2.4 (11.83)

14. Secondary Outcome: Incidence of Clinically Significant Changes in ECG Measurements
Description: To evaluate safety and tolerability of hepatic ultrasound insonification in subjects with T2DM
Time Frame: Screening to Day 28
Measure: Mean (Standard Deviation); unit: clinically significant changes
Arm/Group | Safety Population
Number analyzed (Participants) | 16
clinically significant changes | 0 (0)

15. Secondary Outcome: Change From Baseline in Insulin Sensitivity Index (SI)
Description: To evaluate the effect of hepatic ultrasound insonification on changes from baseline in whole-body insulin sensitivity during a two-step hyperinsulinemic, euglycemic clamp with stable isotope labeled glucose tracer.
  The Insulin Sensitivity Index was to be calculated from the H-E clamp data using the formula included in the SAP, with Step 1 indicating the first phase of the clamp, or the period of administration of the first (lower) insulin infusion rate and Step 2 indicating the second phase of the clamp or the period of administration of the second (higher) insulin infusion rate. Mean GIRs and mean plasma insulin concentrations were to be calculated during steady state for the applicable step(s).
  Change from baseline of SI was then to be computed for each subject as:
  Change from baseline (SI) = SI2 - SI1, where Clamp 2 was the second clamp and Clamp 1 was the first clamp (completed on Day 2, prior to first insonification).
Time Frame: Day 2 (Baseline) to Day 17
Measure: Mean (Standard Deviation); unit: ml/min per microU/ml
Arm/Group | Ultrasound Insonification Effect Population
Number analyzed (Participants) | 14
ml/min per microU/ml | -0.000 (0.0132)

16. Secondary Outcome: Change From Baseline in Glucose Disposal Rate During Steady State (M)
Description: as for outcome 1
Time Frame: Day 2 (Baseline) to Day 17
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Ultrasound Insonification Effect Population
Number analyzed (Participants) | 14
mg/kg/min
  Clamp Timepoint with Low Rate Insulin Infusion (Step 1) | 0.87 (1.623)
  Clamp Timepoint with High Rate Insulin Infusion (Step 2) | 1.04 (3.161)

17. Secondary Outcome: Change From Baseline in Glucose Metabolic Clearance Rate During Steady State (MCR)
Description: as for outcome 1
Time Frame: Day 2 (Baseline) to Day 17
Measure: Mean (Standard Deviation); unit: dL/kg/min
Arm/Group | Ultrasound Insonification Effect Population
Number analyzed (Participants) | 14
dL/kg/min
  Clamp Timepoint with Low Rate Insulin Infusion (Step 1) | 0.81 (1.458)
  Clamp Timepoint with High Rate Insulin Infusion (Step 2) | 0.90 (3.501)

18. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment of Insulin Resistance (HOMA2-IR)
Description: To evaluate the effect of hepatic ultrasound insonification on glucose metabolism parameters, assessed by a Homeostasis Model. A higher value denotes an increased level of insulin resistance, and a lower value denotes an decreased level of insulin resistance. The value is computed based on fasting insulin and glucose values.
  The HOMA2 results were produced by the HOMA2 calculator with FPG and insulin concentration obtained from safety laboratory assessments as the inputs to the calculator at https://www.dtu.ox.ac.uk/homacalculator/. Please see citation (see references module): "Levy 1998 Levy JC, Matthews DR, & Hermans MP. (1998). Correct homeostasis model assessment (HOMA) evaluation uses the computer program. Diabetes Care. 21:2191-2192."
Time Frame: Day 15 (Baseline) to Day 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety Population
Number analyzed (Participants) | 16
score on a scale | -0.81 (1.018)

19. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment of Insulin Secretion (HOMA2-B)
Description: To evaluate the effect of hepatic ultrasound insonification on glucose metabolism parameters, assessed by a Homeostasis Model. The HOMA2 results were to be produced by the HOMA2 calculator with FPG and insulin concentration obtained from safety laboratory assessments as the inputs to the calculator at https://www.dtu.ox.ac.uk/homacalculator/. HOMA2-B values estimate steady state pancreatic beta cell function, as a percent of a normal reference population. See citation: "Levy JC, Matthews DR, & Hermans MP. (1998). Correct homeostasis model assessment (HOMA) evaluation uses the computer program. Diabetes Care. 21:2191-2192."
Time Frame: Day 15 (Baseline) to Day 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety Population
Number analyzed (Participants) | 16
score on a scale | -15.92 (24.132)

20. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: To evaluate the effect of hepatic ultrasound insonification on glucose metabolism parameters, assessed by fasting plasma glucose blood test
Time Frame: Baseline to Day 18 - Baseline was defined as the last non-missing value collected prior to the first on study hepatic ultrasound insonification
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Safety Population
Number analyzed (Participants) | 16
mg/dL | -3.0 (20.87)

21. Secondary Outcome: Change From Baseline in Oral Glucose Tolerance Test (OGTT) Area Under the Curve (AUC 0-180): Glucose
Description: To evaluate the effect of hepatic ultrasound insonification on change from baseline in glucose tolerance and insulin secretion, assessed by an oral glucose tolerance test (OGTT). AUC in this outcome is calculated using the absolute value of glucose measures (compared to incremental AUC below which uses baseline (time 0 glucose) subtracted values).
Time Frame: Day 1 (Baseline) to Day 16
Measure: Mean (Standard Deviation); unit: (mg hr)/dL
Arm/Group | Safety Population
Number analyzed (Participants) | 16
(mg hr)/dL
  Plasma Glucose Total AUC | -2.112 (86.2483)
  Plasma Glucose Incremental AUC | -0.720 (68.7508)

22. Secondary Outcome: Change From Baseline in Oral Glucose Tolerance Test (OGTT) Area Under the Curve (AUC 0-180): Insulin
Description: To evaluate the effect of hepatic ultrasound insonification on change from baseline in glucose tolerance and insulin secretion, assessed by an oral glucose tolerance test (OGTT). AUC in this outcome is calculated using the absolute value of insulin measures (compared to incremental AUC below which uses baseline (time 0 insulin) subtracted values).
Time Frame: Day 1 (Baseline) to Day 16
Measure: Mean (Standard Deviation); unit: (mU hr)/L
Arm/Group | Safety Population
Number analyzed (Participants) | 16
(mU hr)/L
  Insulin Total AUC | 13.580 (32.2072)
  Insulin Incremental AUC | 11.777 (24.1236)

23. Secondary Outcome: Change From Baseline in Continuous Glucose Monitoring System (CGMS): Time in Ranges
Description: To evaluate the effect of hepatic ultrasound insonification on glucose metabolism parameters, assessed by a continuous glucose monitoring system (CGMS)
Time Frame: 14:00 on Day -1 to 22:00 on Day 1 (Baseline) to 14:00 on Day 15 to 22:00 on Day 16 - omitting data collected between a subject's OGTT glucose consumption start time + 180 minutes
Measure: Mean (Standard Deviation); unit: % Time in Ranges
Arm/Group | Safety Population
Number analyzed (Participants) | 16
% Time in Ranges
  Time >250 mg/dL | -1.80 (8.376)
  Time >180 mg/dL | -0.90 (12.869)
  Time 70-180 mg/dL | 0.90 (12.869)
  Time <70 mg/dL | -0.00 (0.000)
  Time <54 mg/dL | -0.00 (0.000)

24. Secondary Outcome: Change From Baseline in Continuous Glucose Monitoring System (CGMS): Average Daily Glucose
Description: as for outcome 23
Time Frame: as for outcome 23
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Safety Population
Number analyzed (Participants) | 16
mg/dL | -4.807 (17.0274)

25. Secondary Outcome: Change From Baseline in Continuous Glucose Monitoring System (CGMS): Blood Glucose Coefficient of Variation
Description: as for outcome 23
Time Frame: as for outcome 23
Measure: Mean (Standard Deviation); unit: % Coefficient of Variation
Arm/Group | Safety Population
Number analyzed (Participants) | 16
% Coefficient of Variation | -1.58 (3.858)

26. Secondary Outcome: Change From Baseline in Continuous Glucose Monitoring System (CGMS): Low/High Blood Glucose Index
Description: To evaluate the effect of hepatic ultrasound insonification on glucose metabolism parameters, assessed by a continuous glucose monitoring system (CGMS)
  To calculate the LBGI and HBGI, the original BG data for each day/period was to be transformed such that it was centered by zero and bound between -sqrt(10) and sqrt(10).
  f(BG,α,β) = [(ln(BG))1.084 - 5.381]*1.509
  The transformed values were then to be input into the BG risk function:
  r(BG) = 10 * f(BG,α,β)2
  The risk of each observation was further to be transformed into two series, risk of low BG series, rl(BG), and risk of high BG series, rh(BG):
  rl(BG) = r(BG) if f(BG) < 0 and 0 otherwise rh(BG) = r(BG) if f(BG) > 0 and 0 otherwise These series were then to be averaged to produce the LBGI and the HBGI as shown in the equations in the SAP.
Time Frame: as for outcome 23
Measure: Mean (Standard Deviation); unit: Blood Glucose Index
Arm/Group | Safety Population
Number analyzed (Participants) | 16
Blood Glucose Index
  Low Blood Glucose Index (LBGI) | -0.02 (0.056)
  High Blood Glucose Index (HBGI) | -0.85 (2.951)

27. Secondary Outcome: Incidence of Adverse Device Effects (ADEs) With a Severity Score of 2: Treatment Emergent Adverse Events (TEAEs) by System Organ Class and Preferred Term
Description: as for outcome 5
Time Frame: Screening to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Population
Number analyzed (Participants) | 16
Participants
  Subjects with at least one Treatment Emergent Adverse Event (TEAE) | 0
  Skin and subcutaneous tissue disorders | 0
  Ecchymosis | 0
  Erythema | 0
  Gastrointestinal disorders | 0
  Abdominal pain | 0
  Dyspepsia | 0
  Vomiting | 0
  General disorders and administration site conditions | 0
  Infusion site hemorrhage | 0
  Vessel puncture site swelling | 0
  Metabolism and nutrition disorders | 0
  Hypoglycaemia | 0
  Nervous system disorders | 0
  Dizziness | 0
  Vascular disorders | 0
  Thrombophlebitis | 0
  Treatment Emergent Adverse Device Effect (TEADE) | 0
  TEADE Related to Study Procedure | 0
  Serious TEADE | 0
  TEADE Leading to Study Discontinuation | 0
  Unanticipated Adverse Device Effect (UADE) | 0

28. Secondary Outcome: Incidence of Adverse Device Effects (ADEs) With a Severity Score of 3: Treatment Emergent Adverse Events (TEAEs) by System Organ Class and Preferred Term
Description: as for outcome 5
Time Frame: Screening to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Population
Number analyzed (Participants) | 16
Participants
  Subjects with at least one Treatment Emergent Adverse Event (TEAE) | 0
  Skin and subcutaneous tissue disorders | 0
  Ecchymosis | 0
  Erythema | 0
  Gastrointestinal disorders | 0
  Abdominal pain | 0
  Dyspepsia | 0
  Vomiting | 0
  General disorders and administration site conditions | 0
  Infusion site hemorrhage | 0
  Vessel puncture site swelling | 0
  Metabolism and nutrition disorders | 0
  Hypoglycaemia | 0
  Nervous system disorders | 0
  Dizziness | 0
  Vascular disorders | 0
  Thrombophlebitis | 0
  Treatment Emergent Adverse Device Effect (TEADE) | 0
  TEADE Related to Study Procedure | 0
  Serious TEADE | 0
  TEADE Leading to Study Discontinuation | 0
  Unanticipated Adverse Device Effect (UADE) | 0

29. Secondary Outcome: Incidence of Adverse Device Effects (ADEs) With a Severity Score of 4: Treatment Emergent Adverse Events (TEAEs) by System Organ Class and Preferred Term
Description: as for outcome 5
Time Frame: Screening to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Population
Number analyzed (Participants) | 16
Participants
  Subjects with at least one Treatment Emergent Adverse Event (TEAE) | 0
  Skin and subcutaneous tissue disorders | 0
  Ecchymosis | 0
  Erythema | 0
  Gastrointestinal disorders | 0
  Abdominal pain | 0
  Dyspepsia | 0
  Vomiting | 0
  General disorders and administration site conditions | 0
  Infusion site hemorrhage | 0
  Vessel puncture site swelling | 0
  Metabolism and nutrition disorders | 0
  Hypoglycaemia | 0
  Nervous system disorders | 0
  Dizziness | 0
  Vascular disorders | 0
  Thrombophlebitis | 0
  Treatment Emergent Adverse Device Effect (TEADE) | 0
  TEADE Related to Study Procedure | 0
  Serious TEADE | 0
  TEADE Leading to Study Discontinuation | 0
  Unanticipated Adverse Device Effect (UADE) | 0

30. Secondary Outcome: Incidence of Adverse Device Effects (ADEs) With a Severity Score of 5: Treatment Emergent Adverse Events (TEAEs) by System Organ Class and Preferred Term
Description: as for outcome 5
Time Frame: Screening to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Population
Number analyzed (Participants) | 16
Participants
  Subjects with at least one Treatment Emergent Adverse Event (TEAE) | 0
  Skin and subcutaneous tissue disorders | 0
  Ecchymosis | 0
  Erythema | 0
  Gastrointestinal disorders | 0
  Abdominal pain | 0
  Dyspepsia | 0
  Vomiting | 0
  General disorders and administration site conditions | 0
  Infusion site hemorrhage | 0
  Vessel puncture site swelling | 0
  Metabolism and nutrition disorders | 0
  Hypoglycaemia | 0
  Nervous system disorders | 0
  Dizziness | 0
  Vascular disorders | 0
  Thrombophlebitis | 0
  Treatment Emergent Adverse Device Effect (TEADE) | 0
  TEADE Related to Study Procedure | 0
  Serious TEADE | 0
  TEADE Leading to Study Discontinuation | 0
  Unanticipated Adverse Device Effect (UADE) | 0

31. Other Pre Specified Outcome: Change From Baseline in Exploratory Biomarkers
Description: To evaluate the effect of hepatic ultrasound insonification on glucose metabolism parameters, as assessed by exploratory markers in blood samples
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Safety Population
Number analyzed (Participants) | 16
ng/L
  Ghrelin | 1.5 (37.05)
  Glucagon | -13.7 (25.17)
  Glucagon-Like Peptide-1 | -26.840 (48.8059)
  Leptin | 2770 (6490)

32. Other Pre Specified Outcome: Change From Baseline in Long-term Glucose Parameters: Fructosamine
Description: To evaluate the effect of hepatic ultrasound insonification on glucose metabolism parameters, as assessed by long-term glucose markers in blood samples
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Safety Population
Number analyzed (Participants) | 16
micromol/L | -17.8 (18.35)

33. Other Pre Specified Outcome: Change From Baseline in Long-term Glucose Parameters: Hemoglobin A1C
Description: as for outcome 32
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: % A1C
Arm/Group | Safety Population
Number analyzed (Participants) | 16
% A1C | -0.11 (0.162)

34. Other Pre Specified Outcome: Change From Baseline in Lipid Metabolism Parameters: Cholesterol and Triglycerides
Description: To evaluate the effect of hepatic ultrasound insonification on glucose metabolism parameters, as assessed by lipid metabolism markers in blood samples
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Safety Population
Number analyzed (Participants) | 16
mg/dL
  Change from Baseline in Cholesterol | -10.9 (17.00)
  Change from Baseline in HDL Cholesterol | -3.9 (4.90)
  Change from Baseline in LDL Cholesterol | -4.9 (14.80)
  Change from Baseline in VLDL Cholesterol | -2.1 (5.34)
  Change from Baseline in Triglycerides | -14.3 (33.12)

35. Other Pre Specified Outcome: Change From Baseline in Lipid Metabolism Parameters: Free Fatty Acids
Description: as for outcome 34
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Safety Population
Number analyzed (Participants) | 16
mEq/L | -0.02 (0.286)

36. Other Pre Specified Outcome: Change From Baseline in Inflammatory Biomarkers: Adiponectin
Description: To evaluate the effect of hepatic ultrasound insonification on glucose metabolism parameters, as assessed by inflammatory biomarkers in blood samples
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Safety Population
Number analyzed (Participants) | 16
mg/L | -0.70 (0.896)

37. Other Pre Specified Outcome: Change From Baseline in Inflammatory Biomarkers: C Reactive Protein
Description: as for outcome 36
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Safety Population
Number analyzed (Participants) | 16
mg/L | -0.1 (1.13)

38. Other Pre Specified Outcome: Change From Baseline in Inflammatory Biomarkers: Interleukin-6
Description: as for outcome 36
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Safety Population
Number analyzed (Participants) | 16
ng/L | 1.29 (1.445)

ADVERSE EVENTS:
Time Frame: Assessing the safety and tolerability profile of hepatic ultrasound insonification in subjects with T2DM was an integral objective of this study; adverse event data was collected for study duration (Screening to Day 28).
Description: TEAE was defined as any undesirable and unintended medical event occurring to a subject from the subject's first hepatic ultrasound insonification until post-treatment follow-up. The skin and subcutaneous tissue disorders, GI disorders, general disorders, metabolism and nutrition disorders, nervous system disorders and vascular disorders were not attributable to the device, as no TEADEs were recorded in the study.
Groups:
- Safety Population: The Safety Population was to consist of all subjects who received at least 1 hepatic ultrasound insonification and included 16 subjects (44.4%).
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 7/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=16)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) — The skin and subcutaneous tissue disorders, GI disorders, general disorders, metabolism and nutrition disorders, nervous system disorders and vascular disorders were not attributable to the device, as no TEADEs were recorded in the study.
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — The skin and subcutaneous tissue disorders, GI disorders, general disorders, metabolism and nutrition disorders, nervous system disorders and vascular disorders were not attributable to the device, as no TEADEs were recorded in the study.
Abdominal pain (Gastrointestinal disorders) | 1 (1) — The skin and subcutaneous tissue disorders, GI disorders, general disorders, metabolism and nutrition disorders, nervous system disorders and vascular disorders were not attributable to the device, as no TEADEs were recorded in the study.
Dyspepsia (Gastrointestinal disorders) | 1 (1) — The skin and subcutaneous tissue disorders, GI disorders, general disorders, metabolism and nutrition disorders, nervous system disorders and vascular disorders were not attributable to the device, as no TEADEs were recorded in the study.
Vomiting (Gastrointestinal disorders) | 1 (1) — The skin and subcutaneous tissue disorders, GI disorders, general disorders, metabolism and nutrition disorders, nervous system disorders and vascular disorders were not attributable to the device, as no TEADEs were recorded in the study.
Infusion site haemorrhage (General disorders) | 1 (1) — The skin and subcutaneous tissue disorders, GI disorders, general disorders, metabolism and nutrition disorders, nervous system disorders and vascular disorders were not attributable to the device, as no TEADEs were recorded in the study.
Vessel puncture site swelling (General disorders) | 1 (1) — The skin and subcutaneous tissue disorders, GI disorders, general disorders, metabolism and nutrition disorders, nervous system disorders and vascular disorders were not attributable to the device, as no TEADEs were recorded in the study.
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) — The skin and subcutaneous tissue disorders, GI disorders, general disorders, metabolism and nutrition disorders, nervous system disorders and vascular disorders were not attributable to the device, as no TEADEs were recorded in the study.
Dizziness (Nervous system disorders) | 1 (1) — The skin and subcutaneous tissue disorders, GI disorders, general disorders, metabolism and nutrition disorders, nervous system disorders and vascular disorders were not attributable to the device, as no TEADEs were recorded in the study.
Thrombophlebitis (Vascular disorders) | 1 (1) — The skin and subcutaneous tissue disorders, GI disorders, general disorders, metabolism and nutrition disorders, nervous system disorders and vascular disorders were not attributable to the device, as no TEADEs were recorded in the study.

LIMITATIONS AND CAVEATS:
The Safety Population consisted of subjects who received hepatic ultrasound insonification and included 16 subjects. The Ultrasound Insonification Effect Population consisted of subjects who received hepatic ultrasound insonification and included 15 subjects. Subject 101-029 had unevaluable data and was excluded from Ultrasound Insonification Effect Population. Subject 101-012 had clamp protocol deviation, and Ultrasound Insonification Effect Population was also analyzed excluding subject.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT04502212/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT04502212/SAP_001.pdf